CLINICAL TRIAL: NCT07346001
Title: Impacts of Prolonged Exposure to Added Sugar Warning Labels on Explicit Weight Bias: a Randomized Controlled Trial
Brief Title: Impacts of Sugar Warnings on Weight Bias
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24-0901b
Record Dates: First submitted 2026-01-06; First posted 2026-01-16 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Nutrition; Diet Interventions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control label (Other)
  Interventions: Behavioral: Control label
- Added sugar warning (Experimental)
  Interventions: Behavioral: Added sugar warning

INTERVENTIONS:
Behavioral: Control label — The control label will display a neutral, square-shaped barcode. Labels will be placed on the front of SSB containers in the experimental store.
  Arms: Control label
Behavioral: Added sugar warning — The added sugar warning will be octagon-shaped and will state "HIGH IN ADDED SUGAR." Warnings will be placed on the front of SSB containers in the experimental store.
  Arms: Added sugar warning

SUMMARY:
This study aims to examine the effects of added sugar warning labels for sugar-sweetened beverages (SSBs) on explicit weight bias and body weight attributional judgements. Participants will be assigned to view either control labels or added sugar warning labels applied on SSBs in an experimental store. Participants will shop for beverages in the store and take a computer survey during four visits to the store, spaced approximately one week apart.

DETAILED DESCRIPTION:
This study aims to determine whether applying added sugar warnings on sugary drinks impacts explicit weight bias and body weight attributional judgements. Approximately 543 adults (ages 18 and older) who have bought at least one SSB in the past week will attend four in-person visits at an experimental store, spaced approximately one week apart. Participants will be randomized to see either neutral control labels or added sugar labels on SSB containers during their visits to the experimental store. At each study visit, participants will shop for beverages in the store and take a computer survey. Explicit weight bias and attribution of responsibility for body weight will be assessed via the computer surveys at the first and last visit.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Bought sugary drinks from a store at least once during the past week
* Willing to attend 4 in-person study appointments

Exclusion Criteria:

• Living in the same household as someone else in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 543 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Explicit weight bias, mean score | Assessed via survey after exposure to intervention (i.e., shopping task) 2 times approximately 4 weeks apart (i.e., in visits 1 and 4)
  Explicit weight bias will be measured by survey through seven items. Items will present participants with pairs of antonyms and ask that they select the box between antonyms that they feel best describes their feelings and beliefs about people with obesity: (1) lazy - hard-working, (2) no will power - has will power, (3) good self - control - poor self-control, (4) active - inactive, (5) self-indulgent - self-sacrificing, (6) dislikes food - likes food, (7) undereats - overeats.
  Response options, which will be presented as 5 boxes between antonyms, will be coded in a categorical 1-5 range, where higher scores represent higher endorsement of a stereotype that contributes to weight bias. Each participant's responses to each item will then be averaged across the seven items to obtain their final score on the outcome in a 1-5 range, where higher scores represent higher explicit weight bias.

SECONDARY OUTCOMES:
Body weight attributional judgements, mean score | Assessed via survey after exposure to intervention (i.e., shopping task) 2 times approximately 4 weeks apart (i.e., in visits 1 and 4).
  Body weight attributional judgements will be measured by survey through two items. Items will ask participants how much they agree with two statements: (1) People with obesity are responsible for their weight; (2) People with obesity are to blame for their weight.
  Response options will be on a 5-point scale from strongly disagree to strongly agree, with higher scores representing higher agreement. Each participant's responses to each item will be averaged to obtain their final score on the outcome in a 1-5 range, where higher scores represent higher attribution of personal responsibility for body weight.

CONTACTS AND LOCATIONS:
Overall Officials: Aline D'Angelo Campos, PhD, MPP, Principal Investigator — University of North Carolina, Chapel Hill

IPD SHARING:
Plan to Share IPD: Yes
The Study Protocol and Statistical Analysis Plan will be shared prior to data collection. After data collection and analysis, a de-identified version of individual participant data and the analytic code will be shared through the Open Science Framework (OSF).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The Study Protocol and statistical analysis plan will be available by February 2026 (prior to data collection). A de-identified version of the data collected and analytic code used will become available after data collection and analysis and will remain available indefinitely.
Access Criteria: Open access.
URL: https://osf.io/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2026-01-27): https://cdn.clinicaltrials.gov/large-docs/01/NCT07346001/Prot_SAP_000.pdf